CLINICAL TRIAL: NCT07355088
Title: Precision Subtyping and Prognostic Study of Heart Failure Based on Multi-Omics Integration and Clinical Indicators: A Prospective Single-Center Cohort Study
Acronym: HF-MultiOmics
Status: Not yet recruiting | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Attending Physician, First Affiliated Hospital of Xinjiang Medical University
Other Study IDs: XJMU-HF-MultiOmics-2025-001
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Chronic Heart Failure; Heart Failure With Reduced Ejection Fraction (HFrEF); Heart Failure With Preserved Ejection Fraction (HFPEF); Heart Failure With Mildly Reduced Ejection Fraction (HFmrEF)
Keywords: Chronic Heart Failure; Multi-omics; Gut-heart axis; SGLT2 inhibitors; Risk prediction model; Epicardial Adipose Tissue; Myocardial Strain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The retained biospecimens include:Venous blood samples (for genome, proteome, and metabolome analysis)、Fecal samples (for gut microbiome analysis).All samples will be stored at -80°C after collection and processing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Heart Failure Patients: Enroll 400 participants meeting 2022 ESC guidelines for chronic heart failure (including HFrEF, HFmrEF, HFpEF). Collect clinical data, multi-omics samples, and imaging indicators at baseline; follow up for 12 months to track outcomes and dynamic changes.
- Healthy Controls: Enroll 200 age/gender-matched participants with no history of cardiovascular disease. Collect baseline clinical data and multi-omics samples for comparative analysis; follow up for 12 months.

SUMMARY:
This is a prospective single-center cohort study conducted at The First Affiliated Hospital of Xinjiang Medical University, aiming to enroll 400 patients with chronic heart failure (including HFrEF, HFmrEF, HFpEF) and 200 healthy controls.We will collect clinical data (e.g., NYHA class, NT-proBNP), multi-omics samples (genome, proteome, metabolome, gut microbiome), and imaging indicators (e.g., EAT density, myocardial strain) from participants at baseline. For patients treated with SGLT2 inhibitors, we will also track dynamic changes in multi-omics during follow-up.The main purpose is to build a composite risk prediction model (integrating multi-omics and clinical indicators) to predict the 1-year composite endpoint (heart failure rehospitalization or all-cause death). Secondary goals include identifying specific molecular profiles related to heart failure phenotypes, exploring the "gut-heart axis" mechanism, and finding early biomarkers for SGLT2 inhibitor response.All participants will be followed up for at least 12 months, and the study will strictly comply with ethical norms and protect the privacy of participants.

DETAILED DESCRIPTION:
This prospective single-center cohort study focuses on chronic heart failure (CHF) patients (HFrEF, HFmrEF, HFpEF) and healthy controls, with the core objective of establishing a precision risk stratification model for CHF via multi-omics-clinical integration.

Study Design & Enrollment Participants: 400 CHF patients (meeting 2022 ESC HF guidelines) and 200 age/gender-matched healthy controls (no cardiovascular disease history). Exclusion criteria include acute decompensated HF, end-stage renal disease, active malignancies, and recent antibiotic use (to avoid gut microbiome interference).

Recruitment: Conducted at The First Affiliated Hospital of Xinjiang Medical University over 12 months; eligible participants will provide written informed consent prior to enrollment.

Data & Sample Collection

Baseline:

Clinical data: NYHA functional class, NT-proBNP, echocardiography (LVEF, LVGLS), cardiac CT (EAT density/volume); Multi-omics samples: Plasma (proteome via Olink, metabolome via LC-MS), blood (genome via microarray), feces (gut microbiome via 16S rRNA sequencing; shotgun metagenomics for 200 patients); Follow-up: 3/6/12-month visits to collect clinical outcomes (rehospitalization, mortality), KCCQ quality-of-life scores, and dynamic multi-omics samples (only for SGLT2 inhibitor-treated patients).

Key Analyses Multi-omics characterization: Identify phenotype-specific molecular signatures (e.g., HFpEF-related metabolic profiles) via differential expression and correlation network analysis; Mechanistic exploration: Link gut microbiome composition to circulating metabolites/inflammatory proteins to clarify the "gut-heart axis" in CHF; Model construction: Integrate multi-omics and clinical/imaging indicators to build 4 prediction models (clinical-only, single-omics, multi-omics, integrated), with validation via Harrell's C-statistic and time-dependent ROC.

Quality Control Biological samples: Labeled with unique IDs, stored at -80°C; Imaging data: Independent review by 2 cardiologists (third-party arbitration for discrepancies); Data management: REDCap platform for electronic data capture; independent Data Monitoring Committee (DMC) reviews progress/safety every 6 months.

ELIGIBILITY:
Inclusion Criteria:(1)For chronic heart failure (CHF) patients:1.Meet the 2022 European Society of Cardiology (ESC) diagnostic criteria for CHF, classified into heart failure with reduced ejection fraction (HFrEF), heart failure with mildly reduced ejection fraction (HFmrEF), and heart failure with preserved ejection fraction (HFpEF) per ESC guidelines;2.Aged 18 to 80 years (inclusive);3.Able to provide written informed consent independently (or via a legal guardian if cognitively impaired, with a Mini-Mental State Examination [MMSE] score ≥ 24).

(2)For healthy controls:1.No history of cardiovascular disease, confirmed by medical history review and baseline echocardiography;2.Aged 18 to 80 years (inclusive), matched 1:2 with CHF patients by age and gender;3.Able to provide written informed consent.

Exclusion Criteria:(1)Acute decompensated heart failure (admitted for acute HF exacerbation within 72 hours prior to enrollment);(2)End-stage renal disease, defined as an estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m² (confirmed by serum creatinine testing);(3)Active malignancies (receiving systemic treatment within 6 months prior to enrollment) or severe systemic diseases (e.g., severe liver failure, active autoimmune diseases);(4)Antibiotic use within 2 weeks prior to enrollment (may interfere with gut microbiome analysis);(5)Inability to complete 12-month follow-up (e.g., planned long-term overseas residence) or provide required biological samples (e.g., venous blood, fecal samples).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolls 2 groups of participants at The First Affiliated Hospital of Xinjiang Medical University:(1)400 patients with chronic heart failure (stratified into HFrEF, HFmrEF, and HFpEF per 2022 ESC criteria), aged 18 to 80 years;(2)200 age- and gender-matched healthy controls (1:2 matching ratio with CHF patients) without a history of cardiovascular disease, aged 18 to 80 years.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
1-Year Composite Endpoint by HF Subtype (Heart Failure Rehospitalization or All-Cause Death) | 12 months
  Occurrence of heart failure-related rehospitalization or all-cause death within 12 months after enrollment, stratified by heart failure subtypes (HFrEF, HFmrEF, HFpEF).Subtype stratification is based on the 2022 ESC HF classification criteria; endpoints are confirmed by the study's clinical endpoint adjudication committee.

SECONDARY OUTCOMES:
1-Year Heart Failure-Related Rehospitalization (Independent Endpoint) | 12 months
  Occurrence of rehospitalization due to worsening heart failure (confirmed by clinical symptoms, NT-proBNP elevation, and echocardiographic changes) within 12 months after enrollment.Rehospitalization is verified by hospital admission records and discharge diagnoses; NT-proBNP and echocardiography data are collected from the hospital's electronic medical record system.

OTHER OUTCOMES:
Identification of Heart Failure Phenotype-Specific Molecular Signatures (Multi-Omics Biomarker Panel) | Baseline
  Screening for subtype-specific molecular markers (differentially expressed genes, signature proteins, characteristic metabolites, and gut microbial taxa) that can distinguish heart failure subtypes (HFrEF, HFmrEF, HFpEF) via baseline multi-omics differential analysis.Multi-omics data are analyzed by bioinformatics tools: PCA for dimensionality reduction, DESeq2/limma for differential expression analysis, WGCNA for co-expression network construction; subtype-specific signatures are validated using ROC curves (AUC ≥ 0.75 is considered a potential biomarker).
Correlation Between Multi-Omics Profiles and Clinical Phenotypes of Heart Failure | Baseline
  Correlation between baseline multi-omics profiles (genome, proteome, metabolome, gut microbiome) of heart failure patients and clinical phenotypes (including NYHA functional class, left ventricular ejection fraction [LVEF], NT-proBNP level, and 6-minute walk distance).Correlation is quantified using statistical methods: Pearson correlation analysis (for continuous variables) or Spearman correlation analysis (for categorical variables); partial least squares regression (PLSR) is used to construct the association model between multi-omics features and clinical phenotypes.
Gut-Heart Axis Mechanistic Correlation: Gut Microbiome Composition vs. Circulating Metabolites/Inflammatory Proteins | Baseline
  Gut microbiome: 16S rRNA gene sequencing (Illumina MiSeq platform)，Circulating metabolites: Liquid chromatography-tandem mass spectrometry (LC-MS/MS)，Inflammatory proteins: Multiplex immunoassay (Luminex platform)Spearman correlation analysis (for microbial relative abundance vs. metabolite/protein concentration)；Mantel test (for overall microbiome composition vs. metabolite/protein profiles).

CONTACTS AND LOCATIONS:
Overall Officials: ailiman mahemut, MD, Study Director — First Affiliated Hospital of Xinjiang Medical University; xiang xie, MD, Study Director — First Affiliated Hospital of Xinjiang Medical University; refukait abuduhalike, MD, Study Chair — First Affiliated Hospital of Xinjiang Medical University; aihaidan abuduwayiti, MD, Study Chair — First Affiliated Hospital of Xinjiang Medical University; li zhao, MD, Study Chair — First Affiliated Hospital of Xinjiang Medical University; yujun guo, MM, Study Chair — First Affiliated Hospital of Xinjiang Medical University; zhiying wen, MM, Study Chair — First Affiliated Hospital of Xinjiang Medical University; yanxiao li, MM, Study Chair — Xinjiang Medical University
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, Urumqi, China

IPD SHARING:
Plan to Share IPD: No
This study involves human genetic resources and sensitive clinical data (including multi-omics profiles and patient follow-up information) of participants. According to the regulations on the management of human genetic resources in China and the informed consent agreement signed with participants (which does not include authorization for IPD sharing with external researchers), the individual participant data (IPD) will not be shared with other researchers to protect the privacy and rights of participants, and to comply with relevant national regulations.

REFERENCES:
- [Background] Obermeyer Z, Emanuel EJ. Predicting the Future - Big Data, Machine Learning, and Clinical Medicine. N Engl J Med. 2016 Sep 29;375(13):1216-9. doi: 10.1056/NEJMp1606181. No abstract available. PMID 27682033
- [Background] Antonopoulos AS, Antoniades C. The role of epicardial adipose tissue in cardiac biology: classic concepts and emerging roles. J Physiol. 2017 Jun 15;595(12):3907-3917. doi: 10.1113/JP273049. Epub 2017 Mar 13. PMID 28191635
- [Background] Medvedofsky D, Kebed K, Laffin L, Stone J, Addetia K, Lang RM, Mor-Avi V. Reproducibility and experience dependence of echocardiographic indices of left ventricular function: Side-by-side comparison of global longitudinal strain and ejection fraction. Echocardiography. 2017 Mar;34(3):365-370. doi: 10.1111/echo.13446. Epub 2017 Feb 9. PMID 28185312
- [Background] Tang WH, Wang Z, Levison BS, Koeth RA, Britt EB, Fu X, Wu Y, Hazen SL. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. N Engl J Med. 2013 Apr 25;368(17):1575-84. doi: 10.1056/NEJMoa1109400. PMID 23614584
- [Background] Cheng ML, Wang CH, Shiao MS, Liu MH, Huang YY, Huang CY, Mao CT, Lin JF, Ho HY, Yang NI. Metabolic disturbances identified in plasma are associated with outcomes in patients with heart failure: diagnostic and prognostic value of metabolomics. J Am Coll Cardiol. 2015 Apr 21;65(15):1509-20. doi: 10.1016/j.jacc.2015.02.018. PMID 25881932
- [Background] Zhang X, Schulz BL, Punyadeera C. The current status of heart failure diagnostic biomarkers. Expert Rev Mol Diagn. 2016;16(4):487-500. doi: 10.1586/14737159.2016.1144474. Epub 2016 Feb 17. PMID 26788983
- [Background] Shah S, Henry A, Roselli C, Lin H, Sveinbjornsson G, Fatemifar G, Hedman AK, Wilk JB, Morley MP, Chaffin MD, Helgadottir A, Verweij N, Dehghan A, Almgren P, Andersson C, Aragam KG, Arnlov J, Backman JD, Biggs ML, Bloom HL, Brandimarto J, Brown MR, Buckbinder L, Carey DJ, Chasman DI, Chen X, Chen X, Chung J, Chutkow W, Cook JP, Delgado GE, Denaxas S, Doney AS, Dorr M, Dudley SC, Dunn ME, Engstrom G, Esko T, Felix SB, Finan C, Ford I, Ghanbari M, Ghasemi S, Giedraitis V, Giulianini F, Gottdiener JS, Gross S, Guethbjartsson DF, Gutmann R, Haggerty CM, van der Harst P, Hyde CL, Ingelsson E, Jukema JW, Kavousi M, Khaw KT, Kleber ME, Kober L, Koekemoer A, Langenberg C, Lind L, Lindgren CM, London B, Lotta LA, Lovering RC, Luan J, Magnusson P, Mahajan A, Margulies KB, Marz W, Melander O, Mordi IR, Morgan T, Morris AD, Morris AP, Morrison AC, Nagle MW, Nelson CP, Niessner A, Niiranen T, O'Donoghue ML, Owens AT, Palmer CNA, Parry HM, Perola M, Portilla-Fernandez E, Psaty BM; Regeneron Genetics Center; Rice KM, Ridker PM, Romaine SPR, Rotter JI, Salo P, Salomaa V, van Setten J, Shalaby AA, Smelser DT, Smith NL, Stender S, Stott DJ, Svensson P, Tammesoo ML, Taylor KD, Teder-Laving M, Teumer A, Thorgeirsson G, Thorsteinsdottir U, Torp-Pedersen C, Trompet S, Tyl B, Uitterlinden AG, Veluchamy A, Volker U, Voors AA, Wang X, Wareham NJ, Waterworth D, Weeke PE, Weiss R, Wiggins KL, Xing H, Yerges-Armstrong LM, Yu B, Zannad F, Zhao JH, Hemingway H, Samani NJ, McMurray JJV, Yang J, Visscher PM, Newton-Cheh C, Malarstig A, Holm H, Lubitz SA, Sattar N, Holmes MV, Cappola TP, Asselbergs FW, Hingorani AD, Kuchenbaecker K, Ellinor PT, Lang CC, Stefansson K, Smith JG, Vasan RS, Swerdlow DI, Lumbers RT. Genome-wide association and Mendelian randomisation analysis provide insights into the pathogenesis of heart failure. Nat Commun. 2020 Jan 9;11(1):163. doi: 10.1038/s41467-019-13690-5. PMID 31919418
- [Background] Ibrahim NE, Januzzi JL Jr. Beyond Natriuretic Peptides for Diagnosis and Management of Heart Failure. Clin Chem. 2017 Jan;63(1):211-222. doi: 10.1373/clinchem.2016.259564. Epub 2016 Oct 10. PMID 28062619
- [Background] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313